# **Child Assent Form**

# in relation to the research project: "Developing Innovative PTSD Treatment for Children: Reconsolidation of Traumatic Memories Protocol<sup>TM</sup> for Children (RTM-C Protocol)"

You are invited to participate in a research game using a psychological method called the RTM Protocol<sup>TM</sup> for Children. It helps children feel better when something scares them. We want to understand whether this method works well for children and how to make it even better.

It is safe. I will help you, explain everything, and support you. You can come with mum, dad, or another trusted adult. You may bring your favourite toy.

#### What will we do?

- We will play and watch cartoons.
- You will create films in your imagination.
- I will help you make your scary memories less frightening.

### What is important to know?

- Everything you say or do will be kept secret. No one else will know without your permission.
- You don't have to tell details of events if you don't want to.
- You can say "stop" at any moment.

## Do you want to try?

| Please circle or tick your answer: |
|---------------------------------------------------------|
| () Yes, I want to take part in this research game. |
| () No, I don't want to take part in this research game. |
| Your name: |
| Your signature or drawing: |